CLINICAL TRIAL: NCT07037160
Title: Effectiveness of Foam Rolling Exercise and Kegel Exercise for Urinary Incontinence in Postpartum Women With Diastasis Recti
Brief Title: Effectiveness of Foam RE and KE for Urinary Incontinence in Postpartum Women With Diastasis Recti
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall20/1008
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kegel exercises (Experimental)
  Interventions: Combination Product: Kegel exercises
- Kegel exercises with Foam Rolling (Experimental)
  Interventions: Combination Product: Kegel exercises with Foam Rolling

INTERVENTIONS:
Combination Product: Kegel exercises — Kegel exercises, also known as pelvic floor exercises, involve contracting and relaxing the muscles of the pelvic floor to strengthen them. These exercises can help improve urinary and fecal continence, potentially enhance sexual function, and are recommended for both men and women.
  Arms: Kegel exercises
Combination Product: Kegel exercises with Foam Rolling — Foam rolling can be a helpful tool to prepare for or complement Kegel exercises by releasing tension in surrounding muscles and improving overall pelvic floor function. Foam rolling can help address tight muscles in the hips and lower back that can contribute to pelvic floor dysfunction. By releasing these tight areas, foam rolling can allow for better engagement and control of the pelvic floor muscles during Kegel exercises.
  Arms: Kegel exercises with Foam Rolling

SUMMARY:
The objective of the study will be to assess the efficacy of foam rolling alone and combination treatment of foam rolling and Kegel exercises in alleviating urinary incontinence among postpartum women with diastasis recti.

The data will be collected from 60 enrolled postpartum females with diastasis recti to evaluate the effectiveness of foam rolling alone compared to foam rolling and Kegel exercises in improving urinary incontinence. The data will be collected using urogenital distress inventory (UDI).

DETAILED DESCRIPTION:
Urinary incontinence is a common issue among postpartum women, often linked to diastasis recti, which weakens core and pelvic floor muscles. Despite its prevalence, effective combined treatment approaches remain limited. Foam rolling may enhance muscle function, while Kegel exercises strengthen the pelvic floor. This study investigates their combined effectiveness in managing urinary incontinence among postpartum women with diastasis recti, compared to Kegel exercises alone.

ELIGIBILITY:
Inclusion Criteria:

* Females with age 20 to 35 years
* Females with vaginal delivery
* Non obese females
* Females diagnosed with diastasis recti and urinary incontinence

Exclusion Criteria:

* Females with mental disorders
* Females who take di-uretic medications
* Females with malignant tumors
* Patients with urinary tract infection
* Patients with a history of pelvic surgery
* Patients with cognitive dysfunction
* Female with gynecological conditions or diseases that may affect the investigation results.

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Urogenital Distress Inventory (UDI-6) | 6 Month
  The Urogenital Distress Inventory (UDI-6) is a questionnaire used to assess the impact of urinary symptoms on a woman's quality of life. It consists of six questions, each with four possible responses ranging from "not at all" to "greatly," and the responses are scored from 0 to 3 respectively. The scores for each question are summed, and then the total is multiplied by 33.3 to scale the score to a range of 0-100. Higher scores indicate a greater degree of distress caused by urinary symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Superior University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No